CLINICAL TRIAL: NCT05582044
Title: The Effect of Lower-body Negative Pressure on Exercise Tolerance and Mechanisms of Dyspnea in Heart Failure With Preserved Ejection Fraction
Brief Title: Exercise Lower-body Negative Pressure in Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Neil Eves, professor, University of British Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H22-01882
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Diastolic Dysfunction; Exercise Intolerance; Dyspnea; Pulmonary Congestion; Pulmonary Hemodynamics
MeSH Terms: conditions — Heart Failure; Dyspnea | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled with randomized repeated measures
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind; participants and outcome assessors are blinded to the intervention until data entry and analysis are completed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heart Failure with Preserved Ejection Fraction (40 Participants) (Experimental): Lower-body negative pressure (-15 and -25 mmHg) and neutral pressure (0 mmHg)
  Interventions: Other: Lower-body Negative Pressure (-25 mmHg); Other: Lower-body Negative Pressure (-15 mmHg); Other: Lower-body Neutral Pressure (0 mmHg)
- Healthy Controls (20 Participants) (Active Comparator): Lower-body negative pressure (-15 and -25 mmHg) and neutral pressure (0 mmHg)
  Interventions: Other: Lower-body Negative Pressure (-25 mmHg); Other: Lower-body Negative Pressure (-15 mmHg); Other: Lower-body Neutral Pressure (0 mmHg)

INTERVENTIONS:
Other: Lower-body Negative Pressure (-25 mmHg) — The LBNP chamber will be sealed at the waist prior to Control measures, and the vacuum system will be activated to coincide with the onset of exercise, applying -25mmHg LBNP.
Other: Lower-body Negative Pressure (-15 mmHg) — The LBNP chamber will be sealed at the waist prior to Control measures, and the vacuum system will be activated to coincide with the onset of exercise, applying -15mmHg LBNP.
Other: Lower-body Neutral Pressure (0 mmHg) — In this placebo trial, the LBNP chamber will be sealed at the waist prior to Control measures, and the vacuum system will be activated to coincide with the onset of exercise, but the chamber will be vented to atmosphere.

SUMMARY:
The heart is a pump that must both fill and empty effectively to move blood; if it cannot move enough, heart failure may ensue. Approximately half of all adults living with heart failure have a form where the heart stiffens, which impairs its ability to fill. This form of heart failure particularly affects females and older adults. When people exercise, extra blood returns to the heart. The healthy heart can easily fill and move this extra blood to the muscles. However, when the heart's ability to fill is impaired, the extra blood can back up and pool in the lungs. Blood pooling in the lungs makes people feel breathless, although the investigators do not fully understand why, and this form of heart failure has a high risk of hospitalization and death, but few effective treatments are available. Exercise is one of the few treatments that works well if enough exercise is performed regularly. However, many people with this form of heart failure can only tolerate a small amount before stopping due to severe breathlessness, which can put them off from exercising regularly.

The study's goal is to help these people perform more exercise. The investigators will use a novel form of stationary cycling with a plastic chamber around the lower body that seals at the waist. The chamber can apply suction to the lower body during exercise which will reduce how much extra blood returns and prevent the heart and lungs from being overloaded. Participants will attend 5 visits, including 3 where they will perform a submaximal exercise test for as many minutes as possible with or without light suction. In each of these tests, the investigators will record how long they exercise and ask them to rate how breathless they feel. The investigators will also study their breathing pattern, using a mouthpiece and pressure sensor, and heart function, using ultrasound imaging.

This work will help adults living with heart failure exercise more and improve their health, and help researchers understand what causes breathlessness and develop new treatments.

DETAILED DESCRIPTION:
Heart failure is a major public health issue, affecting >750,000 Canadians and >6 million Americans. Half of all adults with heart failure have a preserved ejection fraction (HFpEF), where left ventricular (LV) diastolic dysfunction (impaired filling) is a key abnormality. These adults have few treatment options other than diuretics and exercise training, but dyspnea (a subjective experience of breathing discomfort) on exertion is a hallmark of HFpEF that causes anxiety, activity avoidance, and a spiral of deconditioning leading to worsening dyspnea and prognosis. Mechanisms of dyspnea on exertion are not well understood in HFpEF, but marked increases in LV filling pressure occur that are associated with lung congestion and interstitial fluid accumulation, which stimulates intrapulmonary afferents and impairs breathing mechanics. During exercise, venous return to the heart increases. This augments stroke volume in health but may overload the LV with diastolic dysfunction and drive lung congestion in HFpEF. As such, attenuating the increase in venous return during exercise may reduce congestion, alleviate dyspnea, and improve exercise tolerance in HFpEF. This concept has been demonstrated by invasively reducing venous return, but the safety and feasibility of invasive approaches is unclear. Lower-body negative pressure (LBNP) is a novel, safe and effective non-invasive means to attenuate venous return that can be applied during cycle exercise and may provide considerable benefit.

Study Aims

1. To investigate whether LBNP can improve exercise tolerance assessed as the time to exercise limitation (TLIM) during constant work-rate exercise in adults with HFpEF.
2. To investigate whether LBNP can attenuate the sensory and affective dimensions of dyspnea during exercise in HFpEF.

Exploratory: To examine the effects of LBNP on central hemodynamics and breathing mechanics during exercise in HFpEF, to explore their relationship with exercise tolerance and dyspnea, and to investigate sex-related differences in these responses and relationships.

Main Endpoints

Primary: Time to exercise limitation (Tlim) measured in seconds during submaximal constant work-rate exercise.

Secondary: Dyspnea intensity measured in Borg units during submaximal constant work-rate exercise.

Study Design

Prospective, two-group (HFpEF and Control), double-blind cross-over study with randomized repeated-measures

Treatment: Lower-body negative pressure (-15 mmHg or -25 mmHg); Placebo: Lower-body atmospheric pressure (0 mmHg)

Study Visits:

Visit 1 [2.0-2.5 hours]: Screening, Enrolment, Phenotyping, and Baseline Testing including anthropometrics, blood pressure, an echocardiogram, pulmonary function tests, and an incremental cardiopulmonary exercise test with 12-lead electrocardiogram.

Visit 2 [0.5 hours]: Venous blood sample for complete blood count (CBC) and B-type natriuretic peptide (NT-proBNP).

Visits 3-5 [1.0-1.5 hours each]: Submaximal Exercise with or without Lower-body Negative Pressure. Participants will undergo assessments of ventilatory and cardiac function while performing 1 submaximal cycle exercise trial per visit with lower-body pressure applied at 0 mmHg, -15 mmHg, or -25 mmHg.

Statistical Analysis

Statistical analyses will be performed using SPSS Statistics (V.28, IBM Inc). Normality will be assessed by the Kolmogorov-Smirnov test. If all compared groups or conditions approximate a normal distribution, data will be presented as mean ± standard deviation with paired comparisons made using t-tests. Otherwise, data will be presented as median (inter-quartile range) with paired comparisons made using the Mann-Whitney U or Wilcoxon Signed Rank tests. Omnibus testing will be conducted using analysis of variance, the Friedman test, or the Kruskal-Wallis test with significant effects tested post hoc using Bonferroni-adjusted t-tests or Dunn's tests. Categorical variables will be summarized as proportions and between-group comparisons will be made using the χ2 test. A two-tailed p <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria for the HFpEF Group:

* Adults with a clinical diagnosis of HFpEF (LV ejection fraction ≥50%) measured in the year prior to Visit 1 (and confirmed at Visit 1), who are New York Heart Association Functional Class II-III (mild-moderate symptoms), ambulatory, receiving guideline-directed medical therapy unchanged for ≥2 months, and clinically stable for ≥3 months.
* Symptom(s) of heart failure requiring treatment within the year prior to Visit 1
* NT-proBNP >50 pmol/L (sinus rhythm) or >150 pmol/L (atrial fibrillation in year prior)
* Diastolic dysfunction based on at least one of the following echocardiographic findings:

  * Left atrial enlargement (diameter >4 cm or volume index >28 mL/m2); or
  * e' <10 cm/s (lateral) or <8 cm/s (septal), or
  * E/e' >10 (lateral), or >15 (septal)

Inclusion Criteria for the Healthy Control Group:

- Healthy sedentary or recreationally active adults from the community

Exclusion Criteria for the HFpEF Group:

* Any prior measurement demonstrated LV ejection fraction ≤40%
* Primary pulmonary, metabolic, renal, hepatic, neuromuscular, or malignant disease
* Primary pulmonary vascular, complex congenital, or > mild valvular heart disease
* Documented infiltrative cardiomyopathy
* Documented valvular or coronary disease requiring intervention
* Myocarditis, pericardial effusion, acute coronary syndrome, or revascularization in the last 3 months
* Resting seated systolic blood pressure >160 mmHg or <100 mmHg
* Jugular venous pressure >12 cm
* Inferior vena cava >2 cm with no inspiratory collapse, or severe right ventricular dysfunction by echo
* Ambulatory supplemental oxygen
* Current or recent participation in >150 min. per week of moderate intensity exercise
* Current or recent (within the past 6 months) smoking
* Body mass index >35 kg/m2
* Contraindication to exercise or otherwise unable to perform cycle ergometry
* Poor echocardiographic imaging windows

Exclusion Criteria for the Healthy Control Group

* Current or recent participation in >150 min. per week of moderate intensity exercise
* History of any cardiovascular condition or cardioactive drug use
* History of any respiratory condition including asthma
* History of any metabolic condition including diabetes
* Non-sinus rhythm
* Echocardiographic evidence of significant left ventricular hypertrophy, valvular abnormalities, left ventricular ejection fraction <50%, or diastolic dysfunction as described in HFpEF inclusion criteria.
* Seated blood pressure ≥140/90 mmHg
* Any other chronic systemic illness
* Current or recent (within the past 6 months) smoking
* Body mass index >35 kg/m2
* Contraindication to exercise or otherwise unable to perform cycle ergometry
* Poor echocardiographic imaging windows

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to exercise limitation (Tlim) | Within 30 minutes of exercise onset
  Exercise will be performed to exhaustion or symptom limitation, and the Tlim will be recorded at the time of cessation to the second

SECONDARY OUTCOMES:
Dyspnea intensity and unpleasantness | Within 30 minutes of exercise onset
  Participants will be asked to rate their dyspnea intensity and dyspnea unpleasantness each out of 10 using the modified Borg scale. Endpoints will be examined at baseline, exercise limitation, and an 'iso-time' defined as the Tlim of the shortest of the 3 tests.

OTHER OUTCOMES:
Left ventricular stroke volume | Within 30 minutes of exercise onset
  Will be calculated from left ventricular volumes measured by echocardiography
Left ventricular filling pressure | Within 30 minutes of exercise onset
  Will be estimated from measurements of left ventricular tissue and blood flow velocities measured by echocardiography
Dynamic lung compliance | Within 30 minutes of exercise onset
  Will be determined from ventilatory pressure-volume loops

CONTACTS AND LOCATIONS:
Overall Officials: Neil D Eves, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada